CLINICAL TRIAL: NCT05104736
Title: A Phase II, Open-Label Trial of PT-112 in Subjects With Thymoma and Thymic Carcinoma
Brief Title: PT-112 in Subjects With Thymoma and Thymic Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000317; 000317-C
Record Dates: First submitted 2021-11-02; First posted 2021-11-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09-17

CONDITIONS: Thymic Epithelial Tumor; Recurrent Thymoma; Thymic Cancer
Keywords: metallo-pyrophosphate; immunogenic cell death; osteotropism; damage-associated molecular patterns; Peripheral Neuropathy
MeSH Terms: conditions — Thymic epithelial tumor; Thymoma; Thymus Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PT-112 (Experimental): PT-112 will be administered intravenously in 28-day cycles, on Days 1 and 15 at a dose of 360 mg/m2 for cycle 1, and on day 1 at 250mg/m2 for each subsequent cycle, until disease progression, development of intolerable adverse events, or until 8 years after an individual participant has been on study
  Interventions: Drug: PT-112

INTERVENTIONS:
Drug: PT-112 — PT-112 will be administered intravenously in 28-day cycles, on Days 1 and 15 at a dose of 360 mg/m2 for cycle 1, and on day 1 at 250mg/m2 for each subsequent cycle,

SUMMARY:
Background:

There are no approved drugs to treat recurrent thymoma and thymic carcinoma. New therapies are needed for people with these cancers. Researchers want to see if the drug PT-112 can help. PT-112 kills cancer cells. It also helps the body s immune system fight cancer.

Objective:

To see if the study drug PT-112 can cause tumors to shrink.

Eligibility:

People ages 18 and older who have thymoma or thymic cancer and whose disease returned or progressed after treatment with at least one platinum-containing chemotherapy, or who have refused standard treatment.

Design:

Participants will be screened with:

Review of medical history and medications

Physical exam

Blood and urine tests

CT or MRI scans of parts of the body, including the brain

Participants will get PT-112 in 28-day cycles, on days 1 and 15 of of the first cycle and on day 1 of each cycle after that. They will get the drug by infusion through a catheter. The catheter is a small plastic tube put into a vein. On days they receive the drug, participants will have physical exams and blood and urine tests. They will have an ECG to test heart function on day 1 of each cycle.

Participants will have scans every 8 weeks.

Participants may choose to have tumor biopsies on day 1 of cycles 1 and 3. Biopsies may be guided by an ultrasound or CT scan.

Participants will continue treatment as long as they can handle the side effects and their disease does not get worse, for up to 8 years.

Participants will have follow-up visits 2 weeks and 4 weeks after they stop therapy. Then the study team will check on participants every 3 months until 8 years after the participant joined the study.

DETAILED DESCRIPTION:
Background

Platinum-based chemotherapy is the standard of care for advanced unresectable thymic epithelial tumors (TETs). However, more than half of these participants experience disease recurrence and require second-line therapy.

There are no approved drugs for treatment of recurrent thymoma and thymic carcinoma and new therapeutic options are needed for participants who have disease progression on or after platinum-containing therapy.

PT-112, a first-in-class metallo-pyrophosphate conjugate, offers a unique set of properties of both cellular interaction and molecular antitumor mechanisms, including resistance to DNA repair pathways and induction of immunogenic cell death.

PT-112 has been clinically proven to be safe and tolerable and has demonstrated efficacy.

Primary Objectives

To determine the objective response rate (ORR) based on RECIST criteria v1.1 to PT-112 in participants with relapsed or refractory TETs

Eligibility

Participants >= age 18 years with histologically confirmed, unresectable thymoma or thymic carcinoma who have previously been treated with at least one platinum-containing chemotherapy regimen or must have refused cytotoxic chemotherapy.

Participants must have progressive and measurable disease

Adequate renal, hepatic and hematopoietic function

Design

This will be a single-arm, open-label study with two cohorts (cohort 1: thymoma; cohort 2: thymic carcinoma) to determine the clinical activity and safety of PT-112 in participants with relapsed or refractory TETs.

PT-112 will be administered intravenously at a dose of 360 mg/m^2 on days 1 and 15 of cycle 1, and at 250 mg/m^2 on day 1 of each subsequent cycle, until disease progression or development of intolerable adverse events. Each cycle is 28 days.

For participants who develop intolerable toxicity at a dose of 360 mg/m^2, dose reduction will be permitted to 300 mg/m^2 after resolution of adverse events to <= grade 1 or baseline. For participants who develop intolerable toxicity at a dose of 250 mg/m^2, up to two dose reductions will be permitted to 200 mg/m^2 or 150 mg/m^2 after resolution of adverse events to <= grade 1 or baseline.

Toxicity will be assessed every cycle by CTCAE, version 5.0.

Tumor response will be assessed after completion of every other cycle (8 weeks) using RECIST criteria, version 1.1. Additionally, for participants with pleural dissemination tumor response will be assessed using International Thymic Malignancy Interest Group (ITMIG) modified RECIST criteria.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically confirmed thymoma or thymic carcinoma.
* Participants should have received at least one prior line of platinum-based chemotherapy. For participants who have refused cytotoxic chemotherapy, a rationale for refusal to receive standard first-line therapy will be captured in the case report form and the medical record. Progressive disease must be documented prior to study entry and participants must have advanced, unresectable disease that is not amenable to surgical resection.
* Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
* Participants must be aged >=18 years.
* ECOG performance status <=1.
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count >= 1,500/mm3 OR >= 1.5 x 10(9)/L
  * platelets >=100,000/mm3 OR (Bullet) 100 x 10(9)/L
  * hemoglobin >= 9g/dL (may have been transfused, at least 7 days prior)
  * total bilirubin <= 1.5 x the upper limit of normal range (ULN)
  * AST(SGOT)/ALT(SGPT) <= 2.5 x ULN OR <= 5 x ULN for participants with documented metastatic disease to the liver
  * creatinine <= 1.5x ULN OR:
  * creatinine clearance >= 60 mL/min/1.73 m2 calculated by calculated using eGRF in the clinical lab
* Negative serum or urine pregnancy test at screening for individuals of childbearing potential (IOCBP). NOTE: IOCBP is defined as any individual who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. Absence of pregnancy must be demonstrated unless there is proven menopause (age >= 50 years and last menarche >= 3 years, or documented menopausal sex hormone profile, or surgical castration) at screening.
* Participants must not become pregnant or start breast feeding during the study. Breastfeeding should be discontinued if the mother is treated with PT-112.
* Individuals of child-bearing potential and those that can father children with a sexual partner of childbearing potential must use medically effective contraception during the study and for 6 months after the last dose of study medication.
* Participants with previously treated brain or CNS metastases are eligible provided that the participant has recovered from any acute side effects of radiotherapy and does not require treatment with steroids, and any whole brain radiation therapy was completed at least 2 weeks prior to initiation of study therapy.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PT-112. Since there is no definitive list of compounds of similar chemical or biologic composition to PT-112, the principal investigator if in doubt, will report known allergies to the pharmacist to make a determination as to whether it is safe to enroll a participant.
* Concurrent treatment with a non-permitted drug.
* Concurrent anticancer treatment within 14 days before initiation of study therapy (includes radiotherapy; however, palliative bone-directed radiotherapy is permitted).
* Major surgery within 14 days before enrollment (excluding prior diagnostic biopsy).
* Concurrent systemic therapy with immunosuppressive agents within 14 days (or 5 half-lives of a drug, whichever is shorter) before initiation of study therapy.
* Use of hormonal agents for anti-cancer therapy within 14 days before initiation of study therapy; or use of any investigational drug within 14 days before initiation of study therapy.
* History of previous malignant disease within the last 2 years with the following exceptions: basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary or follicular thyroid carcinoma, and non-muscle invasive bladder cancer.
* Active infection requiring systemic therapy or significant acute or chronic infections including, among others:

  * Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
  * Known history of testing positive for HIV or known acquired immunodeficiency syndrome with a detectable viral load. However, participants with HIV who have an undetectable viral load and are on stable doses of Highly Active Antiretroviral Therapy (HAART) can be screened for the study.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 5 Grade > 1) with the exception of, alopecia, sensory neuropathy Grade <= 2 and hearing loss Grade <=2.
* Known alcohol or drug abuse.
* Uncontrolled intercurrent illness including, but not limited to the following:

  * Cardiovascular: SYMPTOMATIC congestive heart failure, unstable angina pectoris or cardiac arrhythmia, either active or within the past 6 months
  * Respiratory: Pneumonitis or Idiopathic pulmonary fibrosis (not radiation-associated fibrosis), either active or within the past 6 months
  * Gastrointestinal: Immune colitis or inflammatory bowel disease, either active or within the past 6 months
  * Hematological: Bleeding diathesis or major bleeding events, either active or within the past 6 months
  * Other: psychiatric illness/social situations that would limit compliance with study requirements, including active suicidal ideation or behavior, either active or within the past 12 months
* Administration of live vaccines within 4 weeks prior to treatment. COVID-19 vaccines are permitted at screening.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | assessed every 8 weeks while on treatment and then every 3 months after that for a maximum of 8 years from the start of study
  best overall response is the best response recorded per RECIST 1.1 criteria, from the start of the treatment until disease progression/recurrence

SECONDARY OUTCOMES:
overall response rate (ORR) based on ITMIG modified RECIST (ITMIG) | start of the treatment until disease progression/recurrence for a maximum of 8 years from the start of study
  best overall response is the best response recorded per ITMIG modified RECIST criteria
overall survival (OS) | during treatment and then every 3 months for a maximum of 8 years from the start of study
  time from the date of start of treatment until death from any cause
progression-free survival (PFS) | assessed every 8 weeks while on treatment and then every 3 months for a maximum of 8 years from the start of study
  time from date of start of treatment until time of disease relapse, disease progression, or death
duration of response (DOR) | assessed every 8 weeks while on treatment and then every 3 months for a maximum of 8 years from the start of study
  time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented
safety of PT-112 | safety data routinely collected from initiation of study therapy through long term follow up
  type, frequency, and grade of events will be collected and reported as assessed per CTCAE criteria, version 5

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000317-C.html